CLINICAL TRIAL: NCT00420927
Title: A Multicenter, Randomized, Double-Period, Double - Blind Study to Determine the Optimal Protocol for Treatment Initiation With Methotrexate and Adalimumab Combination Therapy in Patients With Early Rheumatoid Arthritis (OPTIMA)
Brief Title: Study of the Optimal Protocol for Methotrexate and Adalimumab Combination Therapy in Early Rheumatoid Arthritis
Acronym: OPTIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M06-810; 2006-004139-31 (EudraCT Number)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2011-09-29 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis; Tumor Necrosis Factor Optimization
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- ADA+MTX/PBO+MTX (Arm 1) (Experimental): Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1, MTX monotherapy plus blinded placebo (PBO) during Period 2
  Interventions: Biological: adalimumab; Drug: methotrexate; Biological: placebo
- ADA+MTX/ADA+MTX (Arm2) (Experimental): Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1 and Period 2
  Interventions: Biological: adalimumab; Drug: methotrexate
- ADA+MTX/OL ADA+MTX (Arm 3) (Experimental): Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1, open-label combination therapy with ADA + MTX during Period 2
  Interventions: Biological: adalimumab; Drug: methotrexate
- PBO+MTX/PBO+MTX (Arm 4) (Experimental): Methotrexate (MTX) monotherapy plus blinded placebo (PBO) during Period 1 and Period 2
  Interventions: Drug: methotrexate; Biological: placebo
- PBO+MTX/OL ADA+MTX (Arm 5) (Experimental): Methotrexate (MTX) monotherapy plus blinded placebo (PBO) during Period 1, open-label combination therapy with adalimumab (ADA) and MTX during Period 2.
  Interventions: Biological: adalimumab; Drug: methotrexate; Biological: placebo

INTERVENTIONS:
Biological: adalimumab — Adalimumab 40 mg/0.8 mL prefilled syringe injected subcutaneously (SC) every other week (eow)
  Other Names: Humira; D2E7
  Arms: ADA+MTX/ADA+MTX (Arm2); ADA+MTX/OL ADA+MTX (Arm 3); ADA+MTX/PBO+MTX (Arm 1); PBO+MTX/OL ADA+MTX (Arm 5)
Drug: methotrexate — Methotrexate 2.5 mg tablets administered orally once a week starting at 7.5 mg/week with dose escalation (weekly or every other week) by 2.5 mg intervals to 20 mg/week.
Biological: placebo — Placebo for adalimumab 0.8 mL prefilled syringe injected subcutaneously (SC) every other week (eow)
  Arms: ADA+MTX/PBO+MTX (Arm 1); PBO+MTX/OL ADA+MTX (Arm 5); PBO+MTX/PBO+MTX (Arm 4)

SUMMARY:
This study compared the safety and efficacy of combination therapy with adalimumab plus methotrexate (MTX) to that of MTX monotherapy (i.e., placebo plus MTX) in subjects with early rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This was a 78-week, multicenter, randomized, double-blind, double-treatment period study designed to compare the safety and efficacy of adalimumab and MTX with placebo and MTX in subjects with early RA. Subjects were randomized to receive adalimumab 40 mg every other week (eow) or placebo subcutaneous injections in combination with orally administered MTX for 26 weeks (Period 1). All subjects in all arms received open-label MTX weekly throughout the study (both Period 1 and Period 2).

At Weeks 22 and 26, subjects were assessed for achievement of low disease activity, defined as a DAS28 score below 3.2. DAS28 is a measure of RA disease activity calculated using the number of tender and swollen joints (out of a total of 28), C-reactive protein level (CRP, a blood marker of inflammation), and the patient's global assessment of disease activity (indicated by marking a 10 cm line between very good and very bad). Subjects who achieved low disease activity at Week 22 and 26 in the adalimumab arm at the end of Period 1 were randomized to receive MTX monotherapy (placebo and MTX) or combination therapy (adalimumab and MTX) in a 1:1 ratio for the duration of Period 2 (52 weeks, i.e., to Week 78 of the study). Subjects achieving low disease activity at Week 22 and 26 in the placebo arm (MTX monotherapy) at the end of Period 1 continued to receive MTX monotherapy (and placebo injections in a blinded fashion) for the duration of Period 2. Subjects failing to achieve low disease activity at Week 22 and 26 at the end of Period 1 received open-label combination therapy during Period 2 regardless of treatment assignment in Period 1.

ELIGIBILITY:
Inclusion Criteria

* Subject must be 18 or older and in good health
* Subject must meet the definition of early rheumatoid arthritis (RA) defined by the 1987-revised American College of Rheumatology (ACR) classification criteria and had disease duration of less than 1 year from diagnosis
* Subject must have a Disease Activity Score (DAS28, based on C-reactive protein) greater than 3.2, at least 6 swollen joints out of the 66 assessed, and at least 8 tender joints out of the 68 assessed
* Subject must fulfill at least one of the following three criteria:

  * Rheumatoid factor positive
  * Greater than 1 joint erosion
  * Anti-cyclic citrullinated peptide (CCP) antibody positive.

Exclusion Criteria

* Subject has previously received systemic anti-tumor necrosis factor (TNF) therapy
* Subject has received any biologic or investigational therapy within 6 weeks prior to Baseline
* Subject has been previously treated with more than 2 disease-modifying antirheumatic drugs (DMARDs) or MTX, had been treated with intra-articular or parenteral administration of corticosteroids in preceding 4 weeks, or had undergone joint surgery within the preceding 2 months at joints to be assessed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032 (Actual)
Dates: Start 2006-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, PhD, Study Director — Abbott
Locations (170):
- United States (49):
  - Site Reference ID/Investigator# 4560, Birmingham, Alabama
  - Site Reference ID/Investigator# 4547, Birmingham, Alabama
  - Site Reference ID/Investigator# 6222, Huntsville, Alabama
  - Site Reference ID/Investigator# 4537, Mobile, Alabama
  - Site Reference ID/Investigator# 6758, Tuscaloosa, Alabama
  - Site Reference ID/Investigator# 9323, Hemet, California
  - Site Reference ID/Investigator# 4568, La Jolla, California
  - Site Reference ID/Investigator# 4535, Palm Desert, California
  - Site Reference ID/Investigator# 4571, Santa Monica, California
  - Site Reference ID/Investigator# 9271, Torrance, California
  - Site Reference ID/Investigator# 10746, Victorville, California
  - Site Reference ID/Investigator# 4559, Denver, Colorado
  - Site Reference ID/Investigator# 6229, Aventura, Florida
  - Site Reference ID/Investigator# 10603, Lake Mary, Florida
  - Site Reference ID/Investigator# 9325, Orange Park, Florida
  - Site Reference ID/Investigator# 4550, Palm Harbor, Florida
  - Site Reference ID/Investigator# 4570, Sarasota, Florida
  - Site Reference ID/Investigator# 4601, Tampa, Florida
  - Site Reference ID/Investigator# 4552, Vero Beach, Florida
  - Site Reference ID/Investigator# 10745, Meridian, Idaho
  - Site Reference ID/Investigator# 4548, Chicago, Illinois
  - Site Reference ID/Investigator# 4557, Springfield, Illinois
  - Site Reference ID/Investigator# 4605, Wichita, Kansas
  - Site Reference ID/Investigator# 10741, Wheaton, Maryland
  - Site Reference ID/Investigator# 6417, Fall River, Massachusetts
  - Site Reference ID/Investigator# 4561, Dover, New Hampshire
  - Site Reference ID/Investigator# 11222, Freehold, New Jersey
  - Site Reference ID/Investigator# 6228, Passaic, New Jersey
  - Site Reference ID/Investigator# 4544, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 4534, Orchard Park, New York
  - Site Reference ID/Investigator# 9324, Plainview, New York
  - Site Reference ID/Investigator# 4600, Smithtown, New York
  - Site Reference ID/Investigator# 12821, The Bronx, New York
  - Site Reference ID/Investigator# 4549, Mayfield Village, Ohio
  - Site Reference ID/Investigator# 6227, Bend, Oregon
  - Site Reference ID/Investigator# 4546, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 4564, West Reading, Pennsylvania
  - Site Reference ID/Investigator# 4558, Wexford, Pennsylvania
  - Site Reference ID/Investigator# 4533, Charleston, South Carolina
  - Site Reference ID/Investigator# 7482, Greenville, South Carolina
  - Site Reference ID/Investigator# 10743, Jackson, Tennessee
  - Site Reference ID/Investigator# 4562, Nashville, Tennessee
  - Site Reference ID/Investigator# 4536, Dallas, Texas
  - Site Reference ID/Investigator# 4538, Houston, Texas
  - Site Reference ID/Investigator# 6899, San Antonio, Texas
  - Site Reference ID/Investigator# 6381, Tyler, Texas
  - Site Reference ID/Investigator# 10744, Seattle, Washington
  - Site Reference ID/Investigator# 4545, Glendale, Wisconsin
  - Site Reference ID/Investigator# 4572, Oak Creek, Wisconsin
- Argentina (5):
  - Site Reference ID/Investigator# 3886, Buenos Aires
  - Site Reference ID/Investigator# 3888, Buenos Aires
  - Site Reference ID/Investigator# 6346, Buenos Aires
  - Site Reference ID/Investigator# 3887, Quilmes
  - Site Reference ID/Investigator# 3889, San Miguel de Tucumán
- Australia (3):
  - Site Reference ID/Investigator# 8380, Campsie, Sydney
  - Site Reference ID/Investigator# 6954, Clayton
  - Site Reference ID/Investigator# 6940, Malvern East
- Austria (6):
  - Site Reference ID/Investigator# 3915, Graz
  - Site Reference ID/Investigator# 3911, Graz
  - Site Reference ID/Investigator# 3880, Vienna
  - Site Reference ID/Investigator# 3885, Vienna
  - Site Reference ID/Investigator# 3916, Vienna
  - Site Reference ID/Investigator# 7792, Vienna
- Belgium (7):
  - Site Reference ID/Investigator# 3914, Brussels
  - Site Reference ID/Investigator# 3909, Genk
  - Site Reference ID/Investigator# 3881, Gilly
  - Site Reference ID/Investigator# 3376, Liège
  - Site Reference ID/Investigator# 6720, Mechelen
  - Site Reference ID/Investigator# 6718, Sint-Niklaas
  - Site Reference ID/Investigator# 3910, Yvoir
- Canada (17):
  - Site Reference ID/Investigator# 6701, Burlington
  - Site Reference ID/Investigator# 6834, Edmonton
  - Site Reference ID/Investigator# 7197, Halifax
  - Site Reference ID/Investigator# 3883, Hamilton
  - Site Reference ID/Investigator# 3884, Hamilton
  - Site Reference ID/Investigator# 3907, Montreal
  - Site Reference ID/Investigator# 3903, Montreal
  - Site Reference ID/Investigator# 5178, Ottawa
  - Site Reference ID/Investigator# 3904, Richmond
  - Site Reference ID/Investigator# 3912, Sainte-Foy, Quebec
  - Site Reference ID/Investigator# 3901, Sarnia
  - Site Reference ID/Investigator# 3906, St. John's
  - Site Reference ID/Investigator# 6542, Toronto
  - Site Reference ID/Investigator# 3882, Victoria
  - Site Reference ID/Investigator# 5616, Windsor
  - Site Reference ID/Investigator# 5847, Winnipeg
  - Site Reference ID/Investigator# 3905, Winnipeg
- Czechia (5):
  - Site Reference ID/Investigator# 3968, Brno
  - Site Reference ID/Investigator# 3971, Hradec Králové
  - Site Reference ID/Investigator# 5559, Ostrava
  - Site Reference ID/Investigator# 3969, Prague
  - Site Reference ID/Investigator# 5548, Uherské Hradiště
- France (4):
  - Site Reference ID/Investigator# 3982, Amiens
  - Site Reference ID/Investigator# 3979, Le Mans
  - Site Reference ID/Investigator# 3983, Paris
  - Site Reference ID/Investigator# 3918, Strasbourg
- Germany (14):
  - Site Reference ID/Investigator# 3926, Bad Nauheim
  - Site Reference ID/Investigator# 3928, Buch
  - Site Reference ID/Investigator# 3978, Damp
  - Site Reference ID/Investigator# 3924, Düsseldorf
  - Site Reference ID/Investigator# 3965, Frankfurt
  - Site Reference ID/Investigator# 3927, Frankfurt am Main
  - Site Reference ID/Investigator# 3925, Freiburg im Breisgau
  - Site Reference ID/Investigator# 4291, Halle
  - Site Reference ID/Investigator# 8489, Hofheim
  - Site Reference ID/Investigator# 3923, Munich
  - Site Reference ID/Investigator# 8483, Osnabrück
  - Site Reference ID/Investigator# 8486, Ratingen
  - Site Reference ID/Investigator# 3919, Vogelsang-Gommern
  - Site Reference ID/Investigator# 6637, Zerbst
- Hungary (3):
  - Site Reference ID/Investigator# 3921, Budapest
  - Site Reference ID/Investigator# 3922, Budapest
  - Site Reference ID/Investigator# 3920, Debrecen
- Mexico (7):
  - Site Reference ID/Investigator# 3824, Aguascallentes
  - Site Reference ID/Investigator# 3822, León
  - Site Reference ID/Investigator# 3825, Mexico City
  - Site Reference ID/Investigator# 3951, Mexico City
  - Site Reference ID/Investigator# 3890, Mexico City
  - Site Reference ID/Investigator# 3823, Mexico City
  - Site Reference ID/Investigator# 3891, Mexico City
- Netherlands (2):
  - Site Reference ID/Investigator# 3947, Arnhem
  - Site Reference ID/Investigator# 3948, Hilversum
- New Zealand (4):
  - Site Reference ID/Investigator# 8485, Auckland
  - Site Reference ID/Investigator# 8488, Hamilton
  - Site Reference ID/Investigator# 8496, Timaru
  - Site Reference ID/Investigator# 8511, Wellington
- Norway (5):
  - Site Reference ID/Investigator# 7607, Ålesund
  - Site Reference ID/Investigator# 7935, Kristiansand
  - Site Reference ID/Investigator# 7506, Levanger
  - Site Reference ID/Investigator# 7511, Lillehammer
  - Site Reference ID/Investigator# 7500, Trondheim
- Poland (4):
  - Site Reference ID/Investigator# 3963, Bydgoszcz
  - Site Reference ID/Investigator# 3962, Katowice
  - Site Reference ID/Investigator# 5560, Lublin
  - Site Reference ID/Investigator# 3961, Wroclaw
- Puerto Rico (4):
  - Site Reference ID/Investigator# 3944, Caguas
  - Site Reference ID/Investigator# 3937, Ponce
  - Site Reference ID/Investigator# 3934, San Juan
  - Site Reference ID/Investigator# 3935, San Juan
- Slovakia (2):
  - Site Reference ID/Investigator# 3959, Piešťany
  - Site Reference ID/Investigator# 3960, Piešťany
- South Africa (6):
  - Site Reference ID/Investigator# 7177, Berea, Durban
  - Site Reference ID/Investigator# 7175, Cape Town
  - Site Reference ID/Investigator# 7178, Cape Town
  - Site Reference ID/Investigator# 7176, Port Elizabeth
  - Site Reference ID/Investigator# 7172, Pretoria
  - Site Reference ID/Investigator# 7174, Soweto
- Spain (10):
  - Site Reference ID/Investigator# 3955, A Coruña
  - Site Reference ID/Investigator# 13661, Bilbao
  - Site Reference ID/Investigator# 3930, Elche (Alicante)
  - Site Reference ID/Investigator# 8524, Madrid
  - Site Reference ID/Investigator# 3956, Madrid
  - Site Reference ID/Investigator# 3943, Madrid
  - Site Reference ID/Investigator# 3931, Madrid
  - Site Reference ID/Investigator# 3957, Oviedo
  - Site Reference ID/Investigator# 3954, Santiago de Compostela
  - Site Reference ID/Investigator# 3932, Zaragoza
- Sweden (5):
  - Site Reference ID/Investigator# 4015, Eskilstuna
  - Site Reference ID/Investigator# 3984, Falun
  - Site Reference ID/Investigator# 4016, Malmo
  - Site Reference ID/Investigator# 4014, Stockholm
  - Site Reference ID/Investigator# 4017, Uppsala
- United Kingdom (8):
  - Site Reference ID/Investigator# 4012, Bath
  - Site Reference ID/Investigator# 8495, Huddersfield
  - Site Reference ID/Investigator# 4048, Leeds
  - Site Reference ID/Investigator# 4013, London
  - Site Reference ID/Investigator# 4046, Newcastle upon Tyne
  - Site Reference ID/Investigator# 4047, Oxford
  - Site Reference ID/Investigator# 3985, Southampton
  - Site Reference ID/Investigator# 7977, York

REFERENCES:
- [Derived] Smolen J, Fleischmann R, Aletaha D, Li Y, Zhou Y, Sainsbury I, Galindo IL. Disease activity improvements with optimal discriminatory ability between treatment arms: applicability in early and established rheumatoid arthritis clinical trials. Arthritis Res Ther. 2019 Nov 10;21(1):231. doi: 10.1186/s13075-019-2005-9. PMID 31707982
- [Derived] Smolen JS, van Vollenhoven RF, Florentinus S, Chen S, Suboticki JL, Kavanaugh A. Predictors of disease activity and structural progression after treatment with adalimumab plus methotrexate or continued methotrexate monotherapy in patients with early rheumatoid arthritis and suboptimal response to methotrexate. Ann Rheum Dis. 2018 Nov;77(11):1566-1572. doi: 10.1136/annrheumdis-2018-213502. Epub 2018 Aug 3. PMID 30076156
- [Derived] Kavanaugh A, van Vollenhoven RF, Fleischmann R, Emery P, Sainsbury I, Florentinus S, Chen S, Guerette B, Kupper H, Smolen JS. Testing treat-to-target outcomes with initial methotrexate monotherapy compared with initial tumour necrosis factor inhibitor (adalimumab) plus methotrexate in early rheumatoid arthritis. Ann Rheum Dis. 2018 Feb;77(2):289-292. doi: 10.1136/annrheumdis-2017-211871. Epub 2017 Nov 16. PMID 29146743
- [Derived] Keystone EC, Breedveld FC, van der Heijde D, van Vollenhoven RF, Emery P, Smolen JS, Sainsbury I, Florentinus S, Kupper H, Chen K, Kavanaugh A. Achieving comprehensive disease control in patients with early and established rheumatoid arthritis treated with adalimumab plus methotrexate versus methotrexate alone. RMD Open. 2017 Sep 26;3(2):e000445. doi: 10.1136/rmdopen-2017-000445. eCollection 2017. PMID 29018564
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Smolen JS, Emery P, Fleischmann R, van Vollenhoven RF, Pavelka K, Durez P, Guerette B, Kupper H, Redden L, Arora V, Kavanaugh A. Adjustment of therapy in rheumatoid arthritis on the basis of achievement of stable low disease activity with adalimumab plus methotrexate or methotrexate alone: the randomised controlled OPTIMA trial. Lancet. 2014 Jan 25;383(9914):321-32. doi: 10.1016/S0140-6736(13)61751-1. Epub 2013 Oct 26. PMID 24168956

RESULTS

PARTICIPANT FLOW:
Groups:
- ADA+MTX: Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1
- PBO+MTX: Methotrexate (MTX) monotherapy plus blinded placebo during Period 1
- ADA+MTX/ADA+MTX (Arm 2): Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1 and Period 2
- ADA+MTX/OL ADA+MTX (Arm 3): Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1, open-label combination therapy with ADA and MTX during Period 2
Period: Period 1
Arm/Group | ADA+MTX | PBO+MTX | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Started | 515 | 517 | 0 (This treatment group is not relevant to Period 1.) | 0 (This treatment group is not relevant to Period 1.) | 0 (This treatment group is not relevant to Period 1.) | 0 (This treatment group is not relevant to Period 1.) | 0 (This treatment group is not relevant to Period 1.)
Completed | 466 | 460 | 0 | 0 | 0 | 0 | 0
Not Completed | 49 | 57 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 19 | 15 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of efficacy/Loss of efficacy | 1 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject moved/relocated | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliant with study drug | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization error | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Suspected tuberculosis/positive test | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study site closure | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subject received new diagnosis | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Received wrong treatment/incorrect dose | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to meet entry criteria | 8 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Took prohibited medication | 1 | 3 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | ADA+MTX | PBO+MTX | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Started | 0 (This treatment group is not relevant to Period 2.) | 0 (This treatment group is not relevant to Period 2.) | 102 | 105 | 259 | 112 | 348
Completed | 0 | 0 | 89 | 95 | 216 | 97 | 295
Not Completed | 0 | 0 | 13 | 10 | 43 | 15 | 53
Not completed — Adverse Event | 0 | 0 | 7 | 3 | 17 | 6 | 20
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3 | 11 | 2 | 12
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2 | 6 | 3 | 9
Not completed — Lack of efficacy/Loss of efficacy | 0 | 0 | 2 | 1 | 6 | 2 | 6
Not completed — Received wrong treatment/incorrect dose | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Subject unable to find transportation | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Sponsor decision | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Randomization error | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Noncompliant with study drug | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Methotrexate intolerance | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Took prohibited medication | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PBO+MTX: Methotrexate (MTX) monotherapy plus blinded placebo(PBO) during Period 1
- ADA+MTX/PBO+MTX (Arm 1): Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA)during Period 1, MTX monotherapy plus blinded placebo (PBO) during Period 2
- Total: Total of all reporting groups
Arm/Group | ADA+MTX | PBO+MTX | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5) | Total
Number analyzed (Participants) | 515 | 517 | 0 | 0 | 0 | 0 | 0 | 1032
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  |  |  |  |  | 0
  Between 18 and 65 years | 418 | 431 |  |  |  |  |  | 849
  >=65 years | 97 | 86 |  |  |  |  |  | 183
Age Continuous [Mean (Standard Deviation); unit: years] | 50.7 (14.48) | 50.4 (13.62) |  |  |  |  |  | 50.6 (14.05)
Gender [Number; unit: participants]
  Female | 380 | 382 |  |  |  |  |  | 762
  Male | 135 | 135 |  |  |  |  |  | 270
Region of Enrollment [Number; unit: participants]
  Argentina | 32 | 29 |  |  |  |  |  | 61
  Australia | 5 | 8 |  |  |  |  |  | 13
  Austria | 11 | 12 |  |  |  |  |  | 23
  Belgium | 41 | 40 |  |  |  |  |  | 81
  Canada | 57 | 58 |  |  |  |  |  | 115
  Czech Republic | 22 | 19 |  |  |  |  |  | 41
  France | 4 | 8 |  |  |  |  |  | 12
  Germany | 43 | 41 |  |  |  |  |  | 84
  Hungary | 8 | 10 |  |  |  |  |  | 18
  Mexico | 26 | 27 |  |  |  |  |  | 53
  Netherlands | 0 | 3 |  |  |  |  |  | 3
  New Zealand | 3 | 3 |  |  |  |  |  | 6
  Norway | 4 | 5 |  |  |  |  |  | 9
  Poland | 12 | 9 |  |  |  |  |  | 21
  Slovakia | 6 | 3 |  |  |  |  |  | 9
  South Africa | 31 | 32 |  |  |  |  |  | 63
  Spain | 25 | 30 |  |  |  |  |  | 55
  Sweden | 10 | 11 |  |  |  |  |  | 21
  United Kingdom | 26 | 17 |  |  |  |  |  | 43
  United States | 149 | 152 |  |  |  |  |  | 301

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Low Disease Activity (DAS28 Less Than 3.2) and No Radiographic Progression From Baseline (Change in mTSS Less Than or Equal to 0.5) at Week 78, Arm 2 vs. Arm 4
Description: The Disease Activity Score (DAS28) is calculated using the number of tender and swollen joints (out of 28 counted), C-reactive protein level, and the patient's global assessment of disease activity. The calculated range of DAS28 is 0.49 to 9.07, with scores below 3.2 indicating low disease activity. For the modified Total Sharp score (mTSS), x-rays of hand/wrist and feet joints are scored for erosions (0 to 5) and joint space narrowing (0 to 4). The erosion score and the narrowing score are added to determine the total score, which ranges from 0 (no damage) to 448.
Time Frame: Week 78
Population: The analysis was performed on the ITT Population comprised of all subjects who entered Period 2 and received at least 1 dose of study drug (blinded or open-label) during Period 2. Nonresponder imputation was used for missing data.
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 59 | 73 | 94 | 61 | 129
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.023, Chi-squared; P value is from Pearson's chi-square test

2. Secondary Outcome: Number of Subjects With Low Disease Activity (DAS28 Less Than 3.2) and No Radiographic Progression From Baseline (Change in mTSS Less Than or Equal to 0.5) at Week 78, Arm 2 vs. Arm 1
Description: as for outcome 1
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 59 | 73 | 94 | 61 | 129
Statistical Analysis 1: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.082, Regression, Logistic

3. Secondary Outcome: Number of Subjects With DAS28 Low Disease Activity (DAS28 Less Than 3.2) at Week 78
Description: The Disease Activity Score (DAS28) is calculated using the number of tender and swollen joints (out of 28 counted), C-reactive protein level, and the patient's global assessment of disease activity. The calculated range of DAS28 is 0.49 to 9.07. A DAS28 less than 2.6 indicates clinical remission, DAS28 2.6 to 3.2 indicates low disease activity, DAS28 3.2 to less than 5.1 indicates moderate disease activity, and DAS28 of 5.1 or greater indicates high disease activity.
Time Frame: Week 78
Population: ITT Population, Nonresponder imputation
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 71 | 80 | 108 | 78 | 185
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.280, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.287, Regression, Logistic

4. Secondary Outcome: Number of Subjects With DAS28 Remission (DAS28 Less Than 2.6) at Week 78
Description: as for outcome 3
Time Frame: Week 78
Population: ITT Population, nonresponder imputation
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 57 | 77 | 71 | 66 | 138
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.026, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.009, Regression, Logistic

5. Secondary Outcome: Number of Subjects With No Radiographic Progression (Change From Baseline in mTSS Less Than or Equal to 0.5) at Week 78
Description: For the modified Total Sharp score (mTSS), x-rays of hand/wrist and feet joints are scored for erosions (0 to 5) and joint space narrowing (0 to 4). The erosion score and the narrowing score are added to determine the total score, which ranges from 0 (no damage) to 448. An increase in mTSS from baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Week 78
Population: ITT Population, nonresponder imputation
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 102 | 259 | 112 | 348
Participants | 70 | 84 | 182 | 77 | 220
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.060, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.063, Regression, Logistic

6. Secondary Outcome: Number of Subjects Meeting American College of Rheumatology 20% (ACR20) Response Criteria at Week 78
Description: Subjects were responders if they had greater than or equal to 20% improvement in tender joint count; greater than or equal to 20% improvement in swollen joint count; and greater than or equal to 20% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant (C-reactive protein).
Time Frame: Week 78
Population: ITT Population, nonresponder imputation
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 84 | 89 | 172 | 90 | 257
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.395, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.640, Regression, Logistic

7. Secondary Outcome: Number of Subjects Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Week 78
Description: Subjects were responders if they had: greater than or equal to 50% improvement in tender joint count; greater than or equal to 50% improvement in swollen joint count; and greater than or equal to 50% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant (C-reactive protein).
Time Frame: Week 78
Population: ITT Population, nonresponder imputation
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 72 | 82 | 120 | 78 | 198
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.159, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.217, Regression, Logistic

8. Secondary Outcome: Number of Subjects Meeting American College of Rheumatology 70% (ACR70) Response Criteria at Week 78
Description: Subjects were responders if they had: greater than or equal to 70% improvement in tender joint count; greater than or equal to 70% improvement in swollen joint count; and greater than or equal to 70% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant (C-reactive protein).
Time Frame: Week 78
Population: ITT Population, nonresponder imputation
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 57 | 73 | 78 | 64 | 137
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.060, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.043, Regression, Logistic

9. Secondary Outcome: Change From Baseline in DAS28 Score at Week 78
Description: as for outcome 3
Time Frame: Baseline to Week 78
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Scores on a scale | -3.54 (1.259) | -3.71 (1.134) | -2.70 (1.531) | -3.04 (1.513) | -3.07 (1.486)
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.004, ANCOVA; Analysis of covariance adjusting for baseline
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.049, ANCOVA; Analysis of covariance adjusting for baseline

10. Secondary Outcome: Number of Subjects With Clinical Disease Activity Index (CDAI) Low Disease Activity (CDAI Less Than or Equal to 10) at Week 78
Description: The CDAI is calculated using number of swollen joints (28 joints assessed), number of tender joints (28 joints assessed), patient's global assessment of disease activity, and physician's global assessment of disease activity. Scores range from 0 to 76.0, with a higher score reflecting worsening disease.
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 75 | 84 | 109 | 82 | 195
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.240, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.271, Regression, Logistic

11. Secondary Outcome: Number of Subjects With Simplified Disease Activity Index (SDAI) Low Disease Activity (SDAI Less Than or Equal to 11) at Week 78
Description: The SDAI is calculated using number of swollen joints (28 joints assessed), number of tender joints (28 joints assessed), patient's global assessment of disease activity, physician's global assessment of disease activity, and acute phase reactant (C-reactive protein). Scores range from 0.1 to 86.0, with a higher score reflecting worsening disease.
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 73 | 79 | 106 | 76 | 192
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.230, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.550, Regression, Logistic

12. Secondary Outcome: Number of Subjects With Clinical Disease Activity Index (CDAI) Remission (CDAI Less Than or Equal to 2.8) at Week 78
Description: as for outcome 10
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 47 | 58 | 39 | 54 | 94
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.301, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.188, Regression, Logistic

13. Secondary Outcome: Number of Subjects With Simplified Disease Activity Index (SDAI) Remission (SDAI Less Than or Equal to 3.3) at Week 78
Description: as for outcome 11
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 45 | 55 | 39 | 51 | 92
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.314, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.235, Regression, Logistic

14. Secondary Outcome: Change From Baseline in CDAI Score at Week 78
Description: as for outcome 10
Time Frame: Baseline to Week 78
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Scores on a scale | -33.30 (12.808) | -33.29 (12.964) | -29.06 (16.561) | -27.63 (15.526) | -31.30 (14.769)
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.030, ANCOVA; Analysis of covariance adjusting for baseline
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.403, ANCOVA; Analysis of covariance adjusting for baseline

15. Secondary Outcome: Change From Baseline in SDAI Score at Week 78
Description: as for outcome 11
Time Frame: Baseline to Week 78
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Scores on a scale | -35.61 (13.527) | -35.16 (13.784) | -31.00 (17.856) | -29.30 (17.120) | -33.43 (15.852)
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.036, ANCOVA; Analysis of covariance adjusting for baseline
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.349, ANCOVA; Analysis of covariance adjusting for baseline

16. Secondary Outcome: Change From Baseline in Synovitis Score According to the Rheumatoid Arthritis Magnetic Resonance Imaging (RA MRI) Scoring System (RAMRIS) at Week 78
Description: Synovitis was assessed using high-field magnetic resonance imaging (MRI) of the hand and wrist. Images were read and scored according to the Outcomes Measures in Rheumatology Clinical Trials' Rheumatoid Arthritis MRI Scoring System (OMERACT RAMRIS). Synovitis in the wrist and finger joints in the most affected hand was scored from 0 (normal) to 3 (severe), for a maximum total score of 21.
Time Frame: Baseline to Week 78
Population: The analysis is based on the Primary Analysis Set, a subset of the ITT Analysis Set that includes subjects who participated in the 78-week HF MRI substudy and whose Baseline HF MRI data were collected on or before the first study drug dose. Observed scores are used in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 2 | 4 | 14 | 4 | 13
Scores on a scale | 2.00 (2.121) | -3.38 (2.562) | -3.25 (3.631) | -3.88 (3.351) | -4.27 (4.211)
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.037, ANCOVA; Analysis of covariance adjusting for baseline
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance adjusting for baseline

17. Secondary Outcome: Number of Subjects With No Radiographic Progression (Change From Baseline in mTSS of Less Than or Equal to 0.5) and Normal Function (HAQ-DI Less Than 0.5) at Week 78
Description: In the Health Assessment Questionnaire Disability Index (HAQ-DI), participants rated their ability to perform daily tasks on a scale of 0 (without any difficulty) to 3 (unable to do). A mean score of 0-1 represents mild to moderate functional disability, 1-2 represents moderate to severe, 2-3 severe to very severe disability. For the modified Total Sharp score (mTSS), x-rays of hand/wrist and feet joints are scored for erosions (0 to 5) and joint space narrowing (0 to 4). The erosion score and the narrowing score are added to determine the total score, which ranges from 0 (no damage) to 448.
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 49 | 59 | 65 | 53 | 84
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.192, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.241, Regression, Logistic

18. Secondary Outcome: Number of Subjects With No Radiographic Progression (Change From Baseline in mTSS of Less Than or Equal to 0.5), Normal Function (HAQ-DI Less Than or Equal to 0.5), and ACR70 Response at Week 78
Description: In the Health Assessment Questionnaire Disability Index (HAQ-DI), a score of 0-1 represents mild to moderate, 1-2 moderate to severe, 2-3 severe to very severe disability. The modified Total Sharp score (mTSS) ranges from 0 (no joint damage) to 448 (worst joint damage). American College of Rheumatology 70% (ACR70) response indicates at least 70% improvement in tender and swollen joint counts and at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; HAQ-DI; and C-reactive protein.
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 37 | 56 | 40 | 43 | 67
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.028, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.014, Regression, Logistic

19. Secondary Outcome: Number of Subjects With No Radiographic Progression (Change From Baseline in mTSS of Less Than or Equal to 0.5), Normal Function (HAQ-DI Less Than 0.5), and DAS28 Remission (DAS28 Less Than 2.6) at Week 78
Description: In the Health Assessment Questionnaire Disability Index (HAQ-DI), a score of 0-1 represents mild to moderate, 1-2 moderate to severe, 2-3 severe to very severe disability. The modified Total Sharp score (mTSS) ranges from 0 (no joint damage) to 448 (severe joint damage). The Disease Activity Score (DAS28) ranges from 0.49 to 9.07, with scores less than 2.6 indicating clinical remission.
Time Frame: Week 78
Measure: Number; unit: Participants
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5)
Number analyzed (Participants) | 102 | 105 | 259 | 112 | 348
Participants | 39 | 53 | 38 | 43 | 63
Statistical Analysis 1: Comparison: ADA+MTX/ADA+MTX (Arm 2) vs PBO+MTX/PBO+MTX (Arm 4); Test type: Superiority or Other; p = 0.074, Regression, Logistic
Statistical Analysis 2: Comparison: ADA+MTX/PBO+MTX (Arm 1) vs ADA+MTX/ADA+MTX (Arm 2); Test type: Superiority or Other; p = 0.077, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Adverse events reported during Period 1 (Weeks 0 to 26) are presented by Period 1 treatment group. Adverse events reported during Period 2 (Weeks 26 to 78) are presented by Period 2 treatment arm (Arm 1 through Arm 5).
Groups:
- ADA+MTX/PBO+MTX (Arm 1): Blinded combination ADA+MTX therapy during Period 1 and blinded MTX monotherapy during Period 2
- ADA+MTX/ADA+MTX (Arm 2): Blinded combination ADA+MTX therapy during Period 1 and Period 2
- ADA+MTX/OL ADA+MTX (Arm 3): Blinded combination therapy during Period 1, open-label combination therapy during Period 2
- PBO+MTX/PBO+MTX (Arm 4): Blinded MTX monotherapy during Period 1 and Period 2
- PBO+MTX/OL ADA+MTX (Arm 5): Blinded MTX monotherapy during Period 1, open-label combination therapy during Period 2
- Period 1 ADA+MTX: Combination therapy with methotrexate (MTX) and blinded adalimumab (ADA) during Period 1
- Period 1 PBO+MTX: Combination therapy with methotrexate (MTX) and blinded placebo (PBO) during Period 1
Arm/Group | ADA+MTX/PBO+MTX (Arm 1) | ADA+MTX/ADA+MTX (Arm 2) | ADA+MTX/OL ADA+MTX (Arm 3) | PBO+MTX/PBO+MTX (Arm 4) | PBO+MTX/OL ADA+MTX (Arm 5) | Period 1 ADA+MTX | Period 1 PBO+MTX
Serious Adverse Events (participants affected / at risk) | 11/102 | 12/105 | 18/259 | 9/112 | 32/348 | 37/515 | 32/517
Other Adverse Events (participants affected / at risk) | 28/102 | 38/105 | 106/259 | 44/112 | 134/348 | 149/515 | 128/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADA+MTX/PBO+MTX (Arm 1) (N=102) | ADA+MTX/ADA+MTX (Arm 2) (N=105) | ADA+MTX/OL ADA+MTX (Arm 3) (N=259) | PBO+MTX/PBO+MTX (Arm 4) (N=112) | PBO+MTX/OL ADA+MTX (Arm 5) (N=348) | Period 1 ADA+MTX (N=515) | Period 1 PBO+MTX (N=517)
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Adverse event resulted in death of subject
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Adverse event resulted in death of subject
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Adverse event resulted in death of subject, who also had a fatal adverse event of facial palsy (cause of death possibly cerebrovascular accident)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Adverse event resulted in death of subject, who also had a fatal adverse event of confusional state (cause of death possibly cerebrovascular accident)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 — Adverse event resulted in death of 2 subjects in ADA+MTX group during Period 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Microgenia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micromastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritoneal tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Physical abuse (Social circumstances) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 4 | 1 — Adverse event resulted in death of 1 subject in Arm 5
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Adverse event resulted in death of subject
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADA+MTX/PBO+MTX (Arm 1) (N=102) | ADA+MTX/ADA+MTX (Arm 2) (N=105) | ADA+MTX/OL ADA+MTX (Arm 3) (N=259) | PBO+MTX/PBO+MTX (Arm 4) (N=112) | PBO+MTX/OL ADA+MTX (Arm 5) (N=348) | Period 1 ADA+MTX (N=515) | Period 1 PBO+MTX (N=517)
Alanine aminotransferase increased (Investigations) | 5 | 4 | 16 | 3 | 16 | 11 | 14
Bronchitis (Infections and infestations) | 3 | 2 | 14 | 6 | 19 | 16 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 13 | 4 | 14 | 20 | 18
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 10 | 1 | 15 | 23 | 27
Headache (Nervous system disorders) | 2 | 3 | 9 | 2 | 10 | 26 | 24
Hypertension (Vascular disorders) | 1 | 5 | 6 | 6 | 7 | 18 | 19
Influenza (Infections and infestations) | 3 | 6 | 9 | 3 | 11 | 22 | 12
Nasopharyngitis (Infections and infestations) | 5 | 6 | 23 | 4 | 23 | 34 | 25
Nausea (Gastrointestinal disorders) | 7 | 4 | 15 | 9 | 27 | 60 | 55
Sinusitis (Infections and infestations) | 3 | 2 | 9 | 8 | 19 | 13 | 15
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 29 | 7 | 27 | 35 | 38
Urinary tract infection (Infections and infestations) | 2 | 5 | 12 | 5 | 22 | 25 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any investigator or institution that plans on presenting/publishing results disclosure, should provide written notification to Abbott within 60 days of their presentation/publication. Abbott requests that no presentation/publication will be allowed until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay of any proposed presentation/publication maybe requested if Abbott needs to secure patent or other proprietary protection.